CLINICAL TRIAL: NCT04647266
Title: Proof of Concept for the Development of Clinical or Mixed Prognostic Score of Morbidity After Endoscopic Subcostal Dissection for Colorectal Lesions in Nancy's Hospital Since 2016 to Nowadays
Brief Title: Pronostic Score of Morbidity to Determine Risk of Complications After Endoscopic Submucosal Dissection for Colorectal Lesions
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI285
Record Dates: First submitted 2020-11-23; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Polyp of Colon
Keywords: Endoscopic Submucosal Dissection
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endoscopic submucosal dissection — endoscopic submucosal dissection

SUMMARY:
The mains complications in colo-rectal dissection are the pain, the delayed bleeding and the perforation and represent around 10%.

Currently, the procedure is realized during a hospitalization with not real recommendation about the time of this.

There is currently no score established for the colo-rectal endoscopic submucosal dissection.

* To develop clinical or mixed prognostic score after endoscopic subcostal dissection for colorectal lesions in Nancy's hospital.
* Allow to obtain an estimation of number of patients required for a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering of lesion relevant of endoscopic submucosal dissection treatment:
* Lesions for which en bloc resection with snare EMR is difficult to apply i/LST-NG, particularly LST-NG (PD) ii/ Lesions showing a VI-type pit pattern iii/ Carcinoma with shallow T1 (SM) invasion Large depressed-type tumors iv/ Large protruded-type lesions suspected to be carcinoma
* Mucosal tumors with submucosal fibrosis
* Sporadic tumors in conditions of chronic inflammation such as ulcerative colitis
* Local residual or recurrent early carcinomas after endoscopic resection Local res Les lésions de plus
* Male or female patients aged ≥ 18 years old
* Patients able to fill in questionnaires written in French

Exclusion Criteria:

* Suspicion of deep submucosal cancer by analysis of macroscopic appearance (Paris O-III), vascular pattern and pit pattern (SANO IIIB, KUDO Vn)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient, more than 18 years old with no contra indication of the general anesthesia suffering of lesion relevant of endoscopic submucosal dissection treatment.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
To develop clinical or mixed prognostic score after endoscopic subcostal dissection for colorectal lesions in Nancy's hospital. | From 2016 to 2020

SECONDARY OUTCOMES:
Allow to obtain an estimation of number of patients required for a larger study | From 2016 to 2020

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste CHEVAUX, Study Director — Doctor
Locations (1):
- CHRU Brabois, Nancy, Meurthe ET Moselle, France